CLINICAL TRIAL: NCT03775343
Title: Early Postoperative Cognitive Impairment in Elderly Patients Following Ocular Surgery
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Other Study IDs: 1907/2017
Record Dates: First submitted 2018-10-26; First posted 2018-12-13 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Decline
Keywords: Anesthesia; Postoperative cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Cognitive Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of blood taken before and after intervention, investigating biomarkers for cognitive impairment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General Anesthesia: General anesthesia:
  25 patients older than 65 years, undergoing elective eye surgery under general anesthesia.
  Intervention: neurocognitive testing (Neurocognitive Test Battery) preoperative, 6 and 24 hours postoperative.
  Blood sampling before surgery (baseline), immediately postoperative, 6 and 24 hours after surgery.
  Interventions: Diagnostic Test: Neurocognitive Test Battery; Diagnostic Test: Blood sampling
- Local anesthesia with sedoanalgesia: 25 patients older than 65 years, undergoing elective eye surgery under local anesthesia in combination with sedoanalgesia.
  Intervention: neurocognitive testing (Neurocognitive Test Battery) preoperative, 6 and 24 hours postoperative Blood sampling before surgery (baseline), immediately postoperative, 6 and 24 hours after surgery.
  Interventions: Diagnostic Test: Neurocognitive Test Battery; Diagnostic Test: Blood sampling
- Control Group: 25 patients, not undergoing any operative intervention. To determine a normal reference value of cognitive functions, a group of 25 individuals without an operative intervention will be recruited as a control group.
  Intervention: neurocognitive testing (Neurocognitive Test Battery) at 3 determined time points (0, 6 and 24 hours)
  Interventions: Diagnostic Test: Neurocognitive Test Battery

INTERVENTIONS:
Diagnostic Test: Neurocognitive Test Battery — neurocognitive testing: preoperative(baseline), 6 and 24 hours postoperative.
Diagnostic Test: Blood sampling — Blood sampling before surgery (baseline), immediately postoperative, 6 and 24 hours after surgery, investigating plasma levels of S 100-B, CRP, vitamines, homocysteine and folic acid
  Groups: General Anesthesia; Local anesthesia with sedoanalgesia

SUMMARY:
This project will investigate changes in cognitive function in the early postoperative phase (<24 hours) after minor surgery in patients of older age (≥65 years).

DETAILED DESCRIPTION:
Primary aim of this study is to evaluate changes in cognitive function in the early postoperative phase after minor surgery in patients of older age (≥65 years).

Background: Postoperative cognitive dysfunction can be a serious complication after surgery and is associated with higher mortality.Several studies have demonstrated that major surgery and patients of older age are risk factors for the incidence of cognitive decline in the postoperative phase. Only a few studies investigated the early postoperative changes in cognitive function (< 24 hours) after minor, day case surgeries in older patients (≥65 years), demonstrating a higher incidence than observed ≥1 week after surgery.

Aim of the project: This study aimed to investigate changes in cognitive function after minor surgery in an elderly patient cohort.

It is the effort to plan perioperative care that can reduce the incidence of postoperative cognitive dysfunction in elderly.

Hypothesis: The present study support the hypothesis that changes in cognitive function after ocular surgery will be greater in the general anesthesia group compared to the sedoanalgesia group.

Methods:

The study will be conducted as a single center, prospective, observational controlled trial at the Medical University of Vienna, Austria.

This prospective and observational study involves consecutive elderly patients (≥65 years) undergoing a minor surgery using general anesthesia or local anesthesia with sedoanalgesia. Fifty patients, 65 years and older, scheduled for elective minor ocular surgery and 25 participants as control group without surgical intervention will be recruited.

Enrollees will be divided in 3 groups:

25 patients general anaesthesia (GA), 25 patients sedoanalgesia combined with local anaesthesia (SA) and 25 participants as control group(CO) without surgical intervention.

Anesthesia will be induced in a standardized fashion in both groups (GA,SA). At baseline the performance on neurocognitive testing using the Mini Mental State Examination (MMSE) hast to be ≥24, otherwise participants will be excluded.

The design utilizes prospective serial assessments of cognitive status. The participants will be evaluated preoperatively and postoperatively over 3 time-points (preoperatively, 6 and 24 hours after surgery) using the Neurocognitive Test Battery Vienna (NTBV) for cognitive assessment.

At the same time points blood tests for plasma levels of S 100-B, IL-6, CRP, vitamin B 12, vitamin D, homocysteine and folic acid will be taken.

This project will investigate the correlation between perioperative changes in these serum parameters with neurocognitive outcome in the elderly after minor surgery to explore whether the concentrations of these parameters can be used as predictors of postoperative cognitive dysfunction and to provide reference for postoperative cognitive dysfunction prevention, early detection and timely diagnosis and treatment.

Further purpose of this study is to investigate if there is an association between changes in intraoperative cerebral oxygenation, changes in perioperative blood pressure, depth of anaesthesia and the presence of cognitive deterioration after surgery.

It is the effort to plan perioperative care that can reduce the incidence of postoperative changes in cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 65 and older
2. scheduled to undergo elective ocular surgery
3. American Society of Anesthesiologists class I, II or III
4. MMSE score ≥ 24
5. The people signed informed consent.
6. Expected surgical duration <90 minutes
7. Able to follow study instructions.

Exclusion Criteria:

1. Patients age < 65 years
2. Emergent nature of the ocular surgery
3. American Society of Anesthesiologists class IV
4. MMSE score < 24
5. unsigned informed consent
6. Expected surgical duration >90 minutes
7. Not able to follow study instructions.
8. History of psychiatric or neurologic disorders (epilepsy, trauma, stroke,depressive disorders, hemorrhage, transient ischemic attack
9. Drug or substance abuse history

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 50 patients 65 years and older without any significant mental (MMSE ≥24) or neuropsychiatric disorders scheduled for elective ocular surgery requiring general anaesthesia or sedoanalgesia will be undergoing serial cognitive assessements pre- and postoperatively over 3 time-points.
  To determine a normal reference value of cognitive functions, a group of 25 participants in the same age (≥65 years)and without surgical intervention will be recruited as a control group and undergo serial cognitive assessements over 3 time-points.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Test Battery Vienna (NTBV) | before surgery (baseline) and 24 hours after surgery
  The Neuropsychological Test Battery Vienna (NTBV) ist a cognitive test to assess a broad range of cognitive abilities.(Lehrner J., 2007) It was created to detect cognitive impairment in Alzheimer's Disease (Lehrner J., 2007). The investigators will investigate changes in NTBV between baseline compared to 24 hour after minor surgery using regression based z-score analyses (-1,5 - + 1,5 standard deviation(SD) ; > -1,5 SD indicating a larger decline in cognitive function).

SECONDARY OUTCOMES:
Neuropsychological Test Battery Vienna (NTBV) | before surgery(baseline) and 6 hours after surgery
  The Neuropsychological Test Battery Vienna (NTBV) ist a cognitive test. (Lehrner J., 2007)

OTHER OUTCOMES:
Blood sampling- S100b levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of S100-B protein (µg/L) will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- IL-6 levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Serum levels of interleukin-6 type cytokines (IL-6 (pg/mL)) will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- CRP levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of C-Reactive Protein (CRP) (mg/L)will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- vitamin B12 levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of vitamin B12 (pg/mL) will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- vitamin D levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of vitamin D (ng/ml) will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- homocysteine levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of homocysteine (mcmol/L)will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.
Blood sampling- folic acid levels | before surgery, at the end point of surgery, 6 and 24 hours after surgery
  Blood sampling will be taken at all patients scheduled for elective ocular surgery. Levels of folic acid (µg/L) will be obtained from venous blood samples collected before surgery, at the end point of surgery, 6 and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided

REFERENCES:
- [Background] Lehrner, J.; Maly, J.; Gleiß, A.; Auff, E. & Dal-Bianco, P., Demenzdiagnostik mit Hilfe der Vienna Neuropsychologischen Testbatterie (VNTB): Standardisierung, Normierung und Validierung, Psychol. Österreich, 4, 358-365, 2007.
- [Background] Foki T, Hitzl D, Pirker W, Novak K, Pusswald G, Auff E, Lehrner J. Erratum to: Assessment of individual cognitive changes after deep brain stimulation surgery in Parkinson's disease using the Neuropsychological Test Battery Vienna short version. Wien Klin Wochenschr. 2017 Aug;129(15-16):585-587. doi: 10.1007/s00508-017-1210-2. No abstract available. PMID 28741045
- See also: The Neuropsychological Test Battery Vienna (NTBV) — http://www.researchgate.net/publication/272825680_The_Neuropsychological_Test_Battery_Vienna_NTBV